CLINICAL TRIAL: NCT05539729
Title: Impact of Vancomycin on the Gut Microbiome and Immune Function in Multiple Sclerosis
Brief Title: Vancomycin Study in Multiple Sclerosis (MS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Stephanie K Tankou, Assistant Professor, Neurology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO-22-0462
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: gut microbiome; peripheral immune function; neuroinflammation; gut-brain axis
MeSH Terms: conditions — Multiple Sclerosis; Neuroinflammatory Diseases | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Placebo-controlled blinded trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The research team will be blinded to the treatment group (placebo/vancomycin).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vancomycin (Experimental): 125mg antibiotic taken 4 times daily by mouth
  Interventions: Drug: Vancomycin
- Placebo (Placebo Comparator): Matching placebo taken 4 times daily by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vancomycin — A marketed antibiotic (Study Drug) supplied by Amerisource Bergen, by the Mount Sinai Investigational Drug Services (IDS), and encapsulated in red coating to match the placebo.
  Arms: Vancomycin
Drug: Placebo — Placebo created by the IDS and encapsulated in red coating to match the Study Drug.
  Arms: Placebo

SUMMARY:
The overall goal of this study is to elucidate a mechanism by which vancomycin modulates the gut-brain axis in multiple sclerosis (MS). The gut microbiome plays an important role in autoimmunity, including MS. However, the identity of gut microbes modulating neuroinflammation in MS and their mechanisms of action remain obscure. Hence, here the research team proposes to investigate the effects of vancomycin on the gut microbiota composition, peripheral immune function, and brain MRI lesions in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 - 50
* newly diagnosed MS (2017 McDonald criteria), CIS or RIS patients, who have experienced symptoms no earlier than the past year
* treatment naive
* able to understand the risks, benefits, and alternatives of participation and give meaningful consent

Exclusion Criteria:

* antibiotic use within the past 90 days;
* pre- or probiotic use within past month or corticosteroids use within the past month;
* use of tobacco products within the past 1 month;
* history of treatment with immunosuppressants;
* history of gastroenteritis within the past month or diagnosis with a chronic infectious disease, i.e. hepatitis B, C or HIV;
* pregnancy or less than 6 months postpartum;
* irritable bowel syndrome and other bowel dysfunction such as constipation;
* history of bowel surgery;
* inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, diabetes and any other auto-immune illness;
* diagnosis with another neurological disease, behavioral or psychiatric conditions that would be incompatible with a safe and successful participation in the study (such as severe major depression, schizophrenia and presence of psychotic symptoms);
* eating disorders such as anorexia nervosa, bulimia, or binge eating syndrome;
* travel outside of the country within the past month;
* contraindication to vancomycin including estimated glomerular filtration rate of <60ml/min, impaired hearing or known allergy.
* Contraindication to MRI such as implanted metallic objects

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Changes in abundance of butyrate producing bacteria | Baseline up to 6 weeks
  Changes in abundance of butyrate producing bacteria from baseline treatment up to 6 weeks
Changes in Serum Butyrate levels | Baseline up to 6 weeks
  Changes in serum butyrate level from baseline treatment up to 6 weeks
  Butyrate is a substance that is produce when gut bacteria breaks down food. Butyrate can get into our blood circulation and regulate how our immune cells function.
Changes in number of peripheral T cells | Baseline up to 6 weeks
  Change in frequency of peripheral regulatory T cells baseline treatment up to 6 weeks.
  T cells are a type of lymphocyte. Lymphocytes are a type of white blood cell. They make up part of the immune system. T cells help the body fight diseases or harmful substances, such as bacteria or viruses.

SECONDARY OUTCOMES:
Changes in abundance of short chain fatty acids (SCFAs)-producing bacteria | Baseline and 12 months
  Changes in abundance of SCFA-producing bacteria
Change in stool SCFAs levels | Baseline and 12 months
  Change in stool SCFAs levels
  SCFAs are substance that are produce when gut bacteria breaks down food.
Change in serum SCFAs levels | Baseline and 12 months
  Change in serum SCFAs levels
Change in number of gadolium enhancing brain lesions | Baseline and 12 months
  Change in number gadolium enhancing brain lesions
  A lesion is a brain injury caused by inflammation. Gadolinium is a dye that is used to visualize areas of active inflammation in the brain.
Change in volume of gadolium enhancing brain lesions | Baseline and 12 months
Change in number of new brain lesions | Baseline and 12 months
Change in volume of new brain lesions | Baseline and 12 months
Change in number of total brain lesions | Baseline and 12 months
Change in volume of total brain lesions | Baseline and 12 months
Changes in number of paramagnetic rim lesions | Baseline and 12 months
  Changes in number of paramagnetic rim lesions
  Paramagnetic rim lesions are a type of brain injury found in MS patients.
Changes in volume of paramagnetic rim lesions | Baseline and 12 months
  Changes in volume of paramagnetic rim lesions
Changes in thalamic brain volumes | Baseline and 12 months
  Changes in thalamic brain volumes
Changes in cortical brain volumes | Baseline and 12 months
  Changes in cortical brain volumes
Changes in total brain volumes | Baseline and 12 months
  Changes in total brain volumes

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie K Tankou, MD, Principal Investigator — Icahn School of Medicine
Locations (1):
- Corinne Goldsmith Dickinson Center for Multiple Sclerosis at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The investigator is not developing the product. The study has been exempted from an IND by the FDA, since it entails the off-label use of a marketed drug.